CLINICAL TRIAL: NCT02152748
Title: Analysis of Disease Progression and Treatment-Induced Alterations in Glioblastoma - an Integrative Morphological and Molecular Approach
Brief Title: Disease Progression and Treatment-induced Alterations in Glioblastoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Adelheid Wöhrer, Dr.med.univ et scient.med., Medical University of Vienna
Other Study IDs: KLI 394
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Brain Tumor
Keywords: glioblastoma; morphological and molecular changes; progression; therapy-resistance
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Disease Progression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glioblastoma: The aim of this study is to analyze systematically morphological and molecular changes associated with glioblastoma progression and therapy-resistance in matched pre- and post-therapeutic glioblastoma samples.
  Interventions: Genetic: analyze systematically morphological and molecular changes associated with glioblastoma progression and therapy-resistance

INTERVENTIONS:
Genetic: analyze systematically morphological and molecular changes associated with glioblastoma progression and therapy-resistance

SUMMARY:
Summary of scientific evidence and rationale of this project:

Integrative molecular-genetic approaches have provided important insights in the biology of glioblastoma. It has meanwhile become clear, that glioblastoma is not a single tumor entity but comprises different molecular subtypes, which are associated with a distinct genetic/epigenetic signature and prognosis. Multimodal treatment approaches combining radio- and chemotherapy as well as the recent introduction of novel antiangiogenic agents have resulted in increasing survival times and improved quality-of-life of glioblastoma patients. Yet, despite these intense treatment efforts the therapeutic efficacy in glioblastoma patients is limited, leading in virtually all cases to tumor recurrence and death of the patients.

As only a limited fraction of glioblastoma patients undergo second neurosurgery at tumor recurrence (< 10%), post-therapeutic samples are rare and no systematic, large-scale studies exist, which address post-therapeutic morphological and molecular alterations in glioblastoma tumor tissue. Yet, these data would help to improve the understanding of mechanisms involved in therapy-resistance and tumor progression, to develop new therapeutic approaches and could pave the way for personalized treatment strategies.

DETAILED DESCRIPTION:
Objectives of the project:

The aim of this study is to analyze systematically morphological and molecular changes associated with glioblastoma progression and therapy-resistance in matched pre- and post-therapeutic glioblastoma samples.

The following primary aims will be addressed:

1. Morphological characterisation of changes in a large series of matched glioblastoma tissues pertaining to i. Vascularization and hypoxia-mediated factors ii. Tumor necrosis and chemoradiation-induced necrosis iii. Inflammatory response iv. Tumor cellularity and proliferation v. Tumor cell phenotype after treatment e.g. glial-mesenchymal transition
2. Molecular analyses

   i. Transcriptomic, DNA methylation and genomic profiling will be performed to detect changes in gene expression, methylation and copy number aberrations in post-therapeutic as compared to pre-therapeutic tumor tissue. ii. The relationship between the transcriptomic, DNA methylation and genomic profiles will be analyzed.
3. Exploratory analysis of associations between morphological and molecular changes in a screening set of 30 glioblastoma cases (with available fresh frozen tissues at first and second surgery) and subsequent validation of relevant findings in a larger glioblastoma cohort (150 cases with matched formalin-fixed paraffin-embedded tissues) by appropriate methods including immunohistochemistry, fluorescence-in-situ-hybridization, and sequencing.
4. Special attention will be paid to gender-specific patterns of therapy-related changes and tumor progression.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All newly diagnosed GB patients will be identified in the Austrian population since 2007 - after the current firstline therapy has become standard, in order to warrant a homogenously treated patient cohort. GB patients with multiple resections will be identified.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Morphology- based analysis | 24 months
  Histopathological workup and evaluation
Molecular analysis | 24 months
  Assessment of genomic alterations at DNA-, RNA- and methylation level

CONTACTS AND LOCATIONS:
Overall Officials: Adelheid Wöhrer, MD PhD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University of Vienna, Institute of Neurology, Vienna, Vienna, Austria